CLINICAL TRIAL: NCT07247734
Title: The Effect of Colchicine, on Insulin Sensitivity in Individuals With Type 1 Diabetes and Systemic Low-grade Inflammation: A Randomized, Double-Blind, Placebo-Controlled, Investigator-Initiated Trial
Brief Title: The Effect of Colchicine, on Insulin Sensitivity in Individuals With Type 1 Diabetes and Systemic Low-grade Inflammation
Acronym: INS1GHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asger Lund, MD (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Asger Lund, MD, Ass. Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-522528-29-00
Record Dates: First submitted 2025-09-29; First posted 2025-11-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes; Chronic Inflammation; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Being a cross-over trial, participants will undergo 2 treatment periods: 4 weeks of treatment with daily colchicine and 4 weeks of treatment with placebo. The order of the treatment periods is randomized 1:1. Each treatment period will be interposed by 8 weeks of wash-out period. In the end of each treatment period the insulin sensitivity will be evaluated by a hyperinsulinemic, euglycemic clamp.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine first period, placebo second period (Active Comparator): Colchicine daily for 4 weeks, followed by an 8-week washout period, then placebo for 4 weeks.
  Interventions: Drug: Colchicin 0.5 mg once daily for two weeks, then twice daily for two weeks; Drug: Placebo once daily for two weeks, then twice daily for two weeks
- Placebo first period, colchicine second period (Active Comparator): Placebo for 4 weeks followed by an 8-week washout period, then Colchicine daily for 4 weeks.
  Interventions: Drug: Placebo once daily for two weeks, then twice daily for two weeks; Drug: Colchicine tablet 0.5 mg once-daily for two weeks, then twice daily for two weeks

INTERVENTIONS:
Drug: Colchicin 0.5 mg once daily for two weeks, then twice daily for two weeks — Colchicine treatment in the first period
  Other Names: Colrefuz
  Arms: Colchicine first period, placebo second period
Drug: Placebo once daily for two weeks, then twice daily for two weeks — Placebo treatment in the first period
  Arms: Placebo first period, colchicine second period
Drug: Colchicine tablet 0.5 mg once-daily for two weeks, then twice daily for two weeks — Colchicine treatment in the second period
  Arms: Placebo first period, colchicine second period
Drug: Placebo once daily for two weeks, then twice daily for two weeks — Placebo treatment in the second period
  Arms: Colchicine first period, placebo second period

SUMMARY:
The aim for this clinical trial is to evaluate if colchicine in addition to standard of care improves insulin sensitivity in individuals with type 1 diabetes, systemic low-grade inflammaiton and reduced insulin sensitivity. The insulin sensitivity will be evaluated by a hyperinsulinemic, euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than five years according to World Health Organization criteria and c-peptid <200 pmol/L
* Age 18-80 years
* User of a continuous glucose monitor (CGM) system
* Glycated hemoglobin A1c (HbA1c) 42-75 mmol/mol
* Stable insulin therapy (defined as no change in insulin brand and no newly initiated Continuous subcutaneous insulin infusion (CSII) or Multiple dose injection (MDI) therapy) and, if applicable, stable usage of glucose monitoring technology (e.g., continuous glucose monitor or intermittently scanned continuous glucose monitor) ≥ 3 months with either multiple daily injections or continuous subcutaneous insulin infusion
* Estimated glomerular filtration rate ≥ 60 mL/min/L/1.73 m²
* Estimated glucose disposal rate (eGDR)* < 8 mg/kg/min OR insulin usage of ≥1 IU/kg pr day
* C-reactive protein (CRP) hsCRP ≥ 2 mg/L, (measured by high-sensitivity assay)**

Exclusion Criteria:

* Hypoglycaemia unawareness (inability to register low blood glucose) ad modum Pedersen-Bjergaard, 24 unless the individual uses a continuous glucose monitor with alarm function
* Liver disease with elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal (measured at screening visit with the possibility of one repeat analysis within seven days, and the last measured value as being conclusive)
* History of cirrhosis, chronic active hepatitis, or severe hepatic disease
* Inflammatory bowel disease or chronic diarrhoea
* Pre-existing progressive neuromuscular disease or individuals with creatinine kinase levels > three times the upper limit of normal (measured at screening visit with the possibility of one repeat analysis within a week, and the last measured value as being conclusive)
* Cancer or lymphoproliferative disease unless in complete remission for > 5 years
* Blood dyscrasias (e.g., myelodysplastic syndromes or related haematological disorders)
* Leukocyte cell count < 3.0 X 109/L
* Thrombocyte count < 110 X 109/L
* Immunosuppressive therapy or state of chronic immunodeficiency, including infection with human immunodeficiency virus (HIV)
* Treatment with anti-inflammatory drugs (e.g., non-steroidal anti-inflammatory drugs (NSAID), acetylsalicylic acid (ASA), prednisone) or whole-body topical steroid during the study or within four weeks before study start. Inhaled steroids are allowed. Short term oral NSAID treatment (≤ 3 days) within four weeks before study start or during the study period is allowed. Treatment of ASA is allowed for up to 1000 mg daily.
* Treatment with colchicine within 60 days of screening visit
* Known or suspected hypersensitivity to colchicine
* Treatment with glucose lowering drugs other than insulin (e.g., Glucagon Like Peptide 1 (GLP-1) receptor agonists, metformin, selective sodium glucose cotransporter-2 (SGLT2)-inhibitors) during the study period or within four weeks before study start
* Haemodialysis or peritoneal dialysis therapy (since colchicine cannot be removed by dialysis or exchange transfusion)
* Treatment with a P-glycoprotein inhibitor (e.g., azithromycin and verapamil) or a strong CYP3A4 inhibitor (e.g., clarithromycin and ritonavir)
* Intake of grapefruit juice
* Other concomitant disease or treatment that according to the investigator's assessment makes the individual unsuitable for study participation
* Alcohol/drug abuse (assessed by the investigator)
* Regarding fertile women:

  * A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
  * Sterilised or postmenopausal women (no menses for 12 months without an alternative medical cause) can be included without the human chorionic gonadotrophin (hCG)-testing during the trial period
  * Women who are pregnant, intend to become pregnant, or are breastfeeding will not be included in the study
  * Female of childbearing potential: must use highly effective contraceptives during the trial and three months after the trial. To exclude pregnancy, urine hCG tests are performed in relation to all visits (V1-V5) and to the phone call in the washout period (P2) and there will be instructions to ensure monthly testing three months after the end of the trial.
  * The following contraceptive methods are considered highly effective and thus adequate for study enrolment for females if maintained throughout the study duration and three months after the trial: Combined hormonal contraception associated with inhibition of ovulation (containing estrogen and progestogen administered oral, intravaginal or transdermal). Progestogen-only hormonal contraception associated with inhibition of ovulation (admninistered oral, injectable or implantable). Intrauterine device (IUD). Intrauterine hormone-releasing system. Bilateral tubal occlusion. Vasectomised partner. Sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject).
  * Male participants with partners of childbearing potential: must either use a condom or ensure that their partner uses a highly effective contraceptive method during the trial and six months after the trial.
* Pregnant or nursing women
* Participants unable to speak or understand Danish
* Receipt of any investigational drug within 30 days prior to visit 1
* Simultaneous participation in any other clinical intervention trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
Mean difference in M-value | Four weeks of treatment comparing colchicine to placebo.
  Mean difference in insulin sensitivity is measured by the M-value (glucose infusion rate mg/kg/min) during the last 30 minutes of a 180 minutes hyperinsulinemic euglycemic clamp procedure using insulin infusion rate of 60 mU/m²/min

SECONDARY OUTCOMES:
Mean difference in M-value | After four weeks of placebo/colchicine
  Measured in mg/m²/min. Adjusted to body surface area (BSA)
Mean difference in M-value (adjusted to fat free mass (FFM)) | After four weeks of placebo/colchicine
  Measured in mg/kg FFM/min
Mean difference in Insulin Sensitivity Index (ISI) | After four weeks of placebo/colchicine
  Glucose infusion rate / Plasma insulin in steady state
Mean difference in average daily insulin dosage | During four weeks of placebo/colchicine
  Units/day. Total daily dose, short acting, long acting
Fold difference in Insulin sensitivity by estimated glucose disposal rate (eGDR) | After four weeks of placebo/colchicine
  Ratio. It is calculated using clinical variables such as waist circumference, hypertension status, and HbA1c. Higher eGDR values indicate better insulin sensitivity
Fold difference in fasting serum/plasma concentrations of C-reactive protein (CRP) measured by a high-sensitivity assay (hsCRP) (mg/L) | After four weeks of placebo/colchicine
  Ratio
Fold difference in in fasting serum/plasma concentrations iInterleukin 6 (IL-6) (pg/mL) | After four weeks of placebo/colchicine
  Ratio
Fold difference in in fasting serum/plasma concentrations of tumour necrosis factor alpha (TNF alpha) | After four weeks of placebo/colchicine
  Ratio

OTHER OUTCOMES:
Mean difference in respiratory exchange ratio between basal state and during clamp | After four weeks of placebo/colchicine
  Ratio
Adipocyte tissue biopsies | After four weeks of placebo/colchicine
  Ratio. Fold difference in Adipocyte size, Inflammation, Glucose metabolism, Extracellular matrix, Oxygen consumption, Transcriptomics, Proteomics
Time spent in target blood glucose range (3.9 - 10 mmol/L) evaluated by a continous glucose monitor (CGM) | The last 7 days of each treatment period.
  Measured in % of 24 hours.
Time spent in tight range (3.9 - 7.8 mmol/L) evaluated by a continous glucose monitor (CGM) | The last 7 days of each treatment period.
  Measured in % of 24 hours.
Time spent in hyperglycemia level 1 (10-13.9 mmol/L) evaluated by a continous glucose monitor (CGM) | The last 7 days of each treatment period.
  Measured in % of 24 hours.
Time spent in hyperglycemia level 2 (> 13.9 mmol/L) evaluated by a continous glucose monitor (CGM) | The last 7 days of each treatment period.
  Measured in % of 24 hours.
Time spent in hypoglycemia level 1 (3.0-3.8 mmol/L) evaluated by a continous glucose monitor (CGM) | The last 7 days of each treatment period.
  Measured in % of 24 hours.
Time spent in hypoglycemia level 2 (< 3.0 mmol/L)evaluated by a continous glucose monitor (CGM) | The last 7 days of each treatment period.
  Measured in % of 24 hours.
Change in glycaemic variability assessed as coefficient of variance (CV) | The last 7 days of each treatment period.
  %-point
Change in standard deviation evaluated by a continous glucose monitor (mmol/L) | The last 7 days of each treatment period.
  %-point
Mean difference in Body mass index (BMI) | After four weeks of placebo/colchicine
  kg/m²
Fold difference in waist-hip ratio | ratio
  After four weeks of placebo/colchicine
Mean difference in waist circumference | After four weeks of placebo/colchicine
  Cm
Mean difference in systolic blood pressure | After four weeks of placebo/colchicine
  mmHg
Mean difference in diastolic blood pressure | After four weeks of placebo/colchicine
  mmHg
Mean difference in heart rate | After four weeks of placebo/colchicine
  beats per minute
Fold difference in body composition (fat-free mass, total fat mass, visceral fat mass rating and bone mass) as measured by bioimpedance | After four weeks of placebo/colchicine
  Ratio
Fold difference in fasting serum/plasma concentrations of inflammatory biomarkers | After four weeks of placebo/colchicine
  Ratio. Interleukines and other cytokines
Fold difference in fasting serum/plasma concentrations of total leukocyte count, including neutrophil, lymphocyte, basophil and eosinophil counts (10^9/L) | After four weeks of placebo/colchicine
  Ratio.
Fold difference in fasting serum/plasma concentrations of very low-density lipoprotein (VLDL) cholesterol (mmol/L) | After four weeks of placebo/colchicine
  Ratio.
Fold difference in fasting serum/plasma concentrations of hemoglobin A1c (mmol/mol) | After four weeks of placebo/colchicine
  Ratio
Fold difference in fasting serum/plasma concentrations of insulin (pmol/L) | After four weeks of placebo/colchicine
  Ratio
Fold difference fasting serum/plasma concentrations of C-peptide (pmol/L) | After four weeks of placebo/colchicine
  Ratio
Fold difference in fasting serum/plasma concentrations of glucagon (pmol/L) | After four weeks of placebo/colchicine
  Ratio
Mean difference in resting energy expenditure ratio between basal state and during clamp | After four weeks of placebo/colchicine
  Ratio. Participants undergo indirect calorimetry in the basal state and during the clamp (from 120-150 minutes)
Fold difference in FibroScan®-assessed liver steatosis (dB/m) | After four weeks of placebo/colchicine
  Ratio. Measured before- and after each treatment period.
Fold difference in Fatty Liver Index (FLI, range 0-100; higher scores indicate greater likelihood of fatty liver) | After four weeks of placebo/colchicine Ratio
  Ratio
Fold difference in Fibrosis-4 (FIB-4) score | After four weeks of placebo/colchicine
  Ratio. The Fibrosis-4 score is a non-invasive index used to estimate liver fibrosis. It is calculated using age, aspartate aminotransferase, alanine aminotransferase, and platelet count. Scale range: Typically from 0 to greater than 3.25
Fold difference in fasting coagulability as measured by thromboelastography (TEG) | After four weeks of placebo/colchicine
  Ratio. Measured before and after each treatment period.
Fold difference in fasting serum/plasma concentrations of hormones during the HIE clamp | After four weeks of placebo/colchicine
  Ratio. Insulin, C-peptide and other counter-regulatory hormones
Difference in rate of treatment-emergent AEs | From signed consent form to last clamp day (week 16-18)
  Rate ratio
Difference in rate of serious AEs (SAEs) | From signed consent form to last clamp day (week 16-18)
  Rate ratio
Difference in rate of severe hypoglycaemia (defined as hypoglycaemia with need of external assistance) | From signed consent form to last clamp day (week 16-18)
  Rate ratio
Difference in rate of diabetic ketoacidosis | From signed consent form to last clamp day (week 16-18)
  Rate ratio
Change in diabetes treatment satisfactory questionnaire, status version (DTSQs) (From 0 (min) to 6 (max), higher scores indicate a better outcome ) | At Visit 2 (week 0), Visit 3 (week 4), Visit 4 (week 12) and Visit 5 (week 16)
  %-point
Change in diabetes treatment satisfactory questionnaire, change version (DTSQc) (From -3 (min) to 3 (max), higher scores indicate a better outcome | At Visit 3 (week 4) and Visit 5 (week 16)
  %-point
Change in fasting serum/plasma concentrations of hemoglobin (mmol/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of thrombocytes (10^9/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of albumin (g/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of potassium (mmol/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of sodium (mmol/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of creatinine (umol/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of creatine kinase (U/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of estimated glomerular filtration rate (eGFR) (mL/min/1.73 m2) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of alanine aminotransferase (U/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of aspartate aminotransferase (U/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of bilirubin (umol/L) | After four weeks of placebo/colchicine
  %-point
Change in fasting serum/plasma concentrations of amylase (units/L) | After four weeks of placebo/colchicine
  %-point
Fold difference in fasting serum/plasma concentrations of high-density lipoprotein (HDL) cholesterol (mmol/L) | After four weeks of placebo/colchicine
  Ratio.
Fold difference in fasting serum/plasma concentrations of total cholesterol (mmol/L) | After four weeks of placebo/colchicine
  Ratio.
Fold difference in fasting serum/plasma concentrations of triglycerides (mmol/L) | After four weeks of placebo/colchicine
  Ratio.
in fasting serum/plasma concentrations of lipoprotein (a) (mg/L) | After four weeks of placebo/colchicine
  Ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Asger B Lund, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital, Denmark
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region 2900, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
At this stage, no final decision has been made regarding the sharing of individual participant data (IPD). While sharing de-identified data may contribute to transparency, reproducibility, and collaborative progress in type 1 diabetes and metabolic research, several factors must be considered. These include ethical and legal obligations related to participant confidentiality, the need for appropriate data-use agreements, and institutional policies on data governance. The possibility of sharing IPD will be revisited upon study completion, in alignment with ethical approvals, and journal publication policies.